CLINICAL TRIAL: NCT03693118
Title: Influence of Cognitive Function Software Therapy on the Improvement of Manual Skills in Multiple Sclerosis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the study was completed
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Pawlukowska Wioletta, Study Director: Przemysław Nowacki MD, PhD, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PomeranianMU2018
Record Dates: First submitted 2018-09-25; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis
Keywords: manual therapy; multiple sclerosis; rehabilitation; motor cortex; neuroplasticity
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup1, Grup2 (Experimental)
  Interventions: Behavioral: Reh1,Reh2
- Grup1,Grup2 (Experimental)
  Interventions: Behavioral: Reh1,Reh2

INTERVENTIONS:
Behavioral: Reh1,Reh2 — The initial group comprised 86 subjects including. The Nine Hole Peg Test (NHPT), administered to all of the patients, was used to evaluate the subjects' manual dexterity. The standardized scale enabled obtaining scores of high validity (right: r= 0.984, left: r = 0.993). Having been administered the NHPT test the initial 86-patient group was reduced to a cohort of 40 subjects qualified for the study, who were subsequently randomly divided into two groups - the study and the control - each consisting of 20 subjects. Three times a week the study group received the upper limb treatment by means of the cognitive function platform. They were expected to achieve 96 levels of visuo-motor coordination in 3 months or the treatment was to be terminated. Prior to the first session of the treatment the patients were provided with all relevant instructions and information about the test displayed on the monitor. They could also choose which hand they would start with.

SUMMARY:
Multiple Sclerosis (MS) is a chronic demyelinating disease of the central nervous system leading to the impairment of motor, visual and cognitive functions. A standardized rehabilitation of cognitive functions can be provided by a systematized treatment program devised to improve neurological patients' quality of life. The degree of difficulty of the computerized tasks was adapted to a patient's predispositions and modified once a desirable improvement in the practiced skill has reached.

The aim of the study was to assess the influence of cognitive therapy by means of the cognitive software on manual dexterity in patients with multiple sclerosis. We also attempted to establish whether factors like age, sex and Expanded Disability Status Scale (EDSS) scores contribute to the outcomes of that therapy. All patients enrolled will have a documented history of MS disease prior to study enrollment. The EDSS scores varied between 1.5-4 (mean score 2.1). The Nine Hole Peg Test (NHPT), administered to all of the patients, was used to evaluate the subjects' manual dexterity. Having been administered the NHPT test the initial 86-patient group was reduced to a cohort of 40 subjects qualified for the study, who were subsequently randomly divided into two groups - the study and the control - each consisting of 20 subjects. Three times a week the study group received the upper limb treatment by means of the cognitive function platform. They were expected to achieve 96 levels of visuo-motor coordination in 3 months or the treatment was to be terminated. After completing each task the patient would move on to a higher level of difficulty. Failure meant having to redo that particular task. One training session lasted 20 min., after which the patient could take a break.

Having completed the training each patient was administered the NHPT test again in view of assessing the efficiency of their upper limb. Due to progressive deterioration of health and other factors only 10 patients managed to complete the training.

ELIGIBILITY:
Inclusion criteria:

MS clinically diagnosed based on McDonald's criteria of 2011 The EDSS between 1.5-4; relapsing-remitting form MS;

exclusio criteria Mental disorders, alcoholism, severe vision disorders including diplopia coinciding upper limb therapy

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-01-13 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Hand therapy using cognitive functions in patients with MS | 3 months
  Three times a week the study group received the upper limb treatment by means of the cognitive function platform. They were expected to achieve 96 levels of visuo-motor coordination in 3 months or the treatment was to be terminated. After completing each task the patient would move on to a higher level of difficulty. Failure meant having to redo that particular task. One training session lasted 20 min., after which the patient could take a break.

CONTACTS AND LOCATIONS:
Locations (1):
- Departmen of Neurology, Szczecin, Unii Lubelskiej, Poland